CLINICAL TRIAL: NCT04002375
Title: Posterior Approach for Pectouteropexy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Kazibe Koyuncu, Principal investigator, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KK201906
Record Dates: First submitted 2019-06-25; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Apical Prolapse
Keywords: pectouteropexy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pectouteropexy — The surgical procedure was initiated after adhesiolysis had been performed by opening the peritoneal layer along the round ligament toward the pelvic side wall. Preparation started at the right external iliac vein and was performed in the medial and caudal direction. A segment of area approximately 3- 4 cm2 of the right lateral part of the iliopectineal ligament (Cooper ligament) adjacent to the insertion of the iliopsoas muscle was exposed.The peritoneum of the bladder was dissected, and the anterior parts of the distal uterus were prepared for mesh fixation. The uterus was elevated to the intended tension-free position using the transvaginal probe (POP-Q level 0-1). The mesh was fixed anteriorly to the cervix using four polyester permanent sutures (Ethibond Excel®; Ethicon). Finally, the mesh was covered with peritoneum using a continuous monofilament absorbable suture (Maxon™; Medtronic).

SUMMARY:
Pectouteropexy surgery has lower complication rates compared to other sling operations. Sacrocolpopexy is another common procedure for hanging the uterus. Small bowel obstruction, ileus or defecation problems are observed in percentages ranging from 0.1 to 5%. Mesh placed between sacrum and vagina often causes narrowing of the pelvis, adhesions may occur and traumas may occur in hypogastic nerves. However, presacral bleeding, which is the most feared complication of these operations, is a rare but life-threatening condition. In pectouteropexy, it is located away from the bladder, intestine and hypogastric vessels by placing the iliopectineal ligament laterally and eliminates the risk of presacral hemorrhage.

In pectouteropexy surgery, the mesh is placed anterior to the cervix. The points emphasized in the criticisms about this technique, inadequate support of the posterior compartment mesh placed in anterior in a future pregnancy is a possible cesarean section and the negative effects on the delivery process.

Therefore, a new technique of pectouteropexy surgery to the posterior of the cervix instead of the anterior cervix of the cervix, the sacrouterine ligament to reduce the complications that may occur due to this procedure and this study was planned to increase the effectiveness.

DETAILED DESCRIPTION:
The study was planned prospectively. The research is planned to be conducted between 30.06.2019 and 30.12.2019. Study Kartal İstanbul Prof. Dr. Lütfi Kırdar Training and Research Hospital Department of Obstetrics and Gynecology. Under the responsibility of Prof. Dr. Ahmet Kale, it will be conducted by Kazibe Koyuncu. The study was planned as a pilot study since it was planned to investigate the results of performing the surgical method with the posterior approach instead of the anterior approach and it was calculated that the inclusion of 20 patients would be sufficient. It is planned to include 20 patients between 30-60 years of age who applied to hospital with prolapse complaint and completed fertility request. Patients' symptoms and physical examinations will be recorded in accordance with international standards and questionnaires will be applied to the files in order to make objective evaluation before and after surgery. Pre-and post-operative POP-Q classifications will be recorded in the files, PFDI-20 questionnaire evaluating the severity of prolapse before and after the surgery, and PGI questionnaire evaluating postoperative satisfaction. In the pectouteropexy operation we applied to the patients, the support of the uterus posterior was insufficient in the sling fixation with mesh suture to the anterior and iliopectineal ligaments of the uterine cervix. We aimed to increase the efficiency of the operation by hanging the uterine cervix posterolaterale to the iliopectineal ligament with the anterior uterine cervix in order to get better results with this method, which can be applied more safely and easily than the other sling methods. Consent form is attached.

There are validity-reliability studies of the questionnaires to be used in Turkish.

ELIGIBILITY:
Inclusion Criteria:

* 1. Being between 30-60 years of age 2. To be diagnosed with at least Stage 2 apical prolapse 3. To have completed fertility 4. To be treated with pectouteropexy for the prolapse

Exclusion Criteria:

* 1. Having had previous prolapse surgery 2. To have connective tissue diseases 3. Inable to cooperate

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 1. Being between 30-60 years of age
  2. To be diagnosed with at least Stage 2 apical prolapse
  3. To have completed fertility
Enrollment: 20 (Estimated)
Dates: Start 2019-06-30 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-02-27 (Estimated)

PRIMARY OUTCOMES:
POP-Q assesment | postoperative 1. day
  pelvic organ prolapse quantification system assessment, does not have any maximum or minimum value, it is scored according to the visualization and is used to assess the difference of prolapse objectively

SECONDARY OUTCOMES:
operation satisfaction | postoperative 1month
  operation satisfaction will be assessed via patient global impression of improvement, it is scaled one to seven, one is related to be satisfied with the result of operation and seven is related to not satisfied from the operation results
pain scores | postoperative 1. day
  pain scores will be assessed via visual analog scale questionnaire, it is scaled one to ten, one is related to have a little pain and 10 is related to have a lot of pain

IPD SHARING:
Plan to Share IPD: Undecided